CLINICAL TRIAL: NCT01348074
Title: Phase II Study of Double Versus Single Reinitiation Dose of Warfarin After Interruption for Surgery
Brief Title: Reinitiation of Anticoagulation After Temporary Withdrawal of Vitamin K Antagonist
Acronym: DOSIDO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Sam Schulman, Prof., McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGH20090520
Record Dates: First submitted 2011-05-03; First posted 2011-05-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Atrial Fibrillation; Venous Thromboembolism; Heart Valve Disease; Surgery
Keywords: warfarin; surgery; management; thromboembolism; bleeding
MeSH Terms: conditions — Atrial Fibrillation; Venous Thromboembolism; Heart Valve Diseases; Thromboembolism; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Double dose (Experimental): Re-initiation with warfarin at twice the usual maintenance dose the first 2 days, then maintenance dose.
  Interventions: Drug: Double dose
- Usual maintenance dose (No Intervention): Usual maintenance dose from Day 1, i.e. no postoperative loading dose.

INTERVENTIONS:
Drug: Double dose — For each individual the dose on Day 1 and Day 2 will be twice the one normally taken
  Other Names: Loading dose
  Arms: Double dose

SUMMARY:
It is not known how to best restart warfarin after temporary withdrawal. Participants will be randomized to two groups. Group 1 will restart warfarin at their usual maintenance dose, group 2 will restart warfarin at double their maintenance dose for two days followed by their usual maintenance dose. The main outcome parameter will be the number of patients who are back in therapeutic INR (international normalized ratio) range 4, and 9 days after restarting anticoagulation with warfarin. Thromboembolic and/or bleeding events will be recorded as additional parameters. These data will be collected by a standardized telephone interview at 1 month. In addition, the investigators will evaluate a possible prothrombotic state by measuring the potential of thrombin generation and D-dimers in the subset of patients visiting HHS-General Hospital for their INR tests.

DETAILED DESCRIPTION:
We will investigate if it is feasible to use double maintenance dose for the first two administrations of vitamin K antagonists when these drugs were temporarily interrupted and thus keep the time of an increased risk of thromboembolism and duration of "bridging" at a minimum. The control group will consist of patients who resume vitamin K antagonists at their usual maintenance dose. The aim of the study is to establish how to best restart anticoagulation with vitamin K antagonists after temporal withdrawal of these drugs. The main outcome parameter will be the proportion of patients who are back to a therapeutic international normalized ratio (INR) ratio at certain days after restarting vitamin K antagonists. Two additional parameters will be evaluated: Firstly, bleeding and thromboembolic complications will be reported and secondly, a possible prothrombotic state, measured as an elevation of D-dimer, at the initiation of anticoagulation will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Current treatment with warfarin
* Need for temporary interruption for invasive procedure or surgery

Exclusion Criteria:

* Need for post-operative hospitalization more than one day
* Participation in another clinical trial
* No consent given

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2011-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with INR back in therapeutic range Day 5 or Day 10 | Day 5-10
  Proportion of patients with INR 2.0-3.0 on Day 5 or Day 10 (day of invasive procedure defined as Day 1)

SECONDARY OUTCOMES:
Thromboembolic events | 30 days
  Objectively verified arterial or venous thromboembolic events
Major bleeding events | 30 days
  Defined by the ISTH criteria of 2010
Minor bleeding events | 30 days
  Any bleeding requiring medical attention but not fulfilling the criteria of Major bleeding
Laboratory parameters of hypercoagulability | 10 days
  Quantitative D-dimer and Thrombin Generation performed in a subset at day of procedure, day 5 and 10 to identify abnormal rise.

CONTACTS AND LOCATIONS:
Overall Officials: Sam Schulman, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- Thrombosis Service, HHS- General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schulman S, El Bouazzaoui B, Eikelboom JW, Zondag M. Clinical factors influencing the sensitivity to warfarin when restarted after surgery. J Intern Med. 2008 Apr;263(4):412-9. doi: 10.1111/j.1365-2796.2007.01913.x. Epub 2008 Jan 16. PMID 18205763
- [Result] Schulman S, Hwang HG, Eikelboom JW, Kearon C, Pai M, Delaney J. Loading dose vs. maintenance dose of warfarin for reinitiation after invasive procedures: a randomized trial. J Thromb Haemost. 2014 Aug;12(8):1254-9. doi: 10.1111/jth.12613. Epub 2014 Jun 25. PMID 24837794